CLINICAL TRIAL: NCT04878120
Title: Hybrid Closed-Loop Control With Prandial Insulin Dosing Informed by Insulin Sensitivity in Adolescents With Type 1 Diabetes
Brief Title: Hybrid Closed-Loop Control With Smart Prandial Insulin Dosing in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Chiara Fabris, PhD, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 210112; 4-CDA-2020-948-A-N (Other Grant/Funding Number: JDRF International (JDRF))
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Sensitivity (SI); Adolescent; Insulin Pump; Continuous Glucose Monitor (CGM); Hybrid Closed Loop (HCL); Diabetes Camp
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standard HCL System - HCL System with Smart Bolus Calculator (Other): Use of standard HCL system followed by use of HCL system with smart bolus calculator informed by insulin sensitivity
  Interventions: Device: Standard HCL System; Device: HCL System with Smart Bolus Calculator
- HCL System with Smart Bolus Calculator - Standard HCL System (Other): Use of HCL system with smart bolus calculator informed by insulin sensitivity followed by use of standard HCL system
  Interventions: Device: Standard HCL System; Device: HCL System with Smart Bolus Calculator

INTERVENTIONS:
Device: Standard HCL System — Standard HCL system (USS Virginia)
Device: HCL System with Smart Bolus Calculator — HCL system (USS Virginia) with smart bolus calculator informed by insulin sensitivity

SUMMARY:
The objective of this study is to evaluate the safety and feasibility of a smart bolus calculator that adjusts insulin dosing for meals according to real-time insulin sensitivity (SI) in adolescents with type 1 diabetes (T1D) using a hybrid closed loop (HCL) system during an active week of diabetes camp.

DETAILED DESCRIPTION:
This is a single center, double-blind, randomized, crossover trial. The study team will target enrollment of 30 adolescents (age 12 - <18 years) with T1D who currently manage their diabetes with an insulin pump and a continuous glucose monitoring (CGM) system. Participants will be randomized 1:1 to the use of the standard HCL system (USS Virginia) vs. the HCL system with the smart bolus calculator first. The trial will be held at a local camp facility and will consist of EITHER a weeklong (6 day/5 night) camp OR two long weekends (4 day/3 night) separated by a washout period of about one week.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥12 and <18 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of T1D for at least one year
3. Currently using insulin for at least six months
4. Currently using an insulin pump for at least three months
5. Currently using a CGM system for at least three months
6. Having at least 75% of CGM data over the previous four weeks
7. Using insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
8. Access to internet and willingness to upload data during the study as needed
9. For females, not currently known to be pregnant or breastfeeding
10. A negative urine pregnancy test will be required for all females of childbearing potential
11. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
12. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study
13. Total daily insulin dose (TDD) of at least 10 U/day
14. Willingness not to start any non-insulin glucose-lowering agent during the course of the trial (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, biguanides, sulfonylureas and naturaceuticals)
15. Willingness to eat at least 40 grams of carbohydrates per meal
16. An understanding and willingness to follow the protocol and signed informed consent
17. Participants and parent/legal guardians will be proficient in reading and writing in English
18. Willingness to comply with COVID-19 precautions as defined by the study team
19. Having completed a COVID-19 vaccination with an FDA-approved COVID-19 vaccine at least two weeks before the first study admission, and willing to provide a copy of the COVID-19 vaccination card

Exclusion Criteria:

1. Hemoglobin A1c <5% or >10% if measured at screening or available from historical medical report performed within the last 6 months; in absence of a valid HbA1c measurement, average blood glucose estimated from CGM data to be approximately between 100 and 240 mg/dL
2. History of diabetic ketoacidosis (DKA) in the 6 months prior to enrollment
3. Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment
4. Pregnancy or intent to become pregnant during the trial
5. Currently breastfeeding or planning to breastfeed
6. Currently being treated for a seizure disorder
7. Planned surgery during study duration
8. History of cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted)
9. Treatment with any non-insulin glucose-lowering agent (metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals)
10. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
11. Use of an insulin delivery mechanism that is not downloadable by the participant or study team
12. Known contact with COVID-positive individual within 14 days of any study admission without negative follow-up COVID-19 Polymerase Chain Reaction (PCR) test performed 3-5 days after the date of exposure
13. Symptoms of COVID-19 (e.g., fever, shortness of breath, unexpected loss of taste or smell) developed within 14 days of any study admission
14. A positive COVID-19 test within 14 days of any study admission or during study admission participation
15. Not being fully vaccinated at the time of the first camp admission (according to Center for Disease Control (CDC) guidelines a person is intended to be fully vaccinated after two weeks from either the second dose of the Pfizer or Moderna vaccine, or the single dose of the Johnson & Johnson vaccine)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Fabris, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HCL Control With Smart Bolus Calculator - Standard HCL Control: Use of HCL system with smart bolus calculator informed by insulin sensitivity followed by use of standard HCL system
  Standard HCL System: Standard HCL system (USS Virginia)
  HCL System with Smart Bolus Calculator: HCL system (USS Virginia) with smart bolus calculator informed by insulin sensitivity
Period: Overall Study
Arm/Group | Standard HCL System - HCL System With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control
Started | 13 | 12
Completed | 12 | 11
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard HCL Control - HCL Control With Smart Bolus Calculator: Use of standard HCL system followed by use of HCL system with smart bolus calculator informed by insulin sensitivity
- HCL Control With Smart Bolus Calculator - Standard HCL Control: Use of HCL system with smart bolus calculator informed by insulin sensitivity followed by use of standard HCL system
- Total: Total of all reporting groups
Arm/Group | Standard HCL Control - HCL Control With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 11 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.7) | 14.6 (1.3) | 14.2 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 9 | 20
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 7.2 (0.4) | 7.2 (0.8) | 7.2 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Low Blood Glucose Index (LBGI)
Description: LBGI computed from CGM collected in the four hours following the dinner meal.
  LBGI is a metric quantifying the risk for hypoglycemia (the higher the LBGI, the higher the exposure to/risk of hypoglycemia), calculated based on the following two steps:
  1. Transforming each CGM reading in the time-series of length N into a hypoglycemia risk score (rL(i), i=1,...,N) by applying the following transformation:
     rL(i) = 10 x (1.509 x (log(CGM(i))^1.084 - 5.381))^2, if CGM(i) <=112.5 mg/dL; rL(i) = 0, if CGM(i) >112.5 mg/dL
  2. Averaging the risk scores rL(i), i=1,...,N.
  The hypoglycemia risk score ranges from 0 for CGM readings >112.5 mg/dL (no hypoglycemia risk) to 100 for CGM readings =20 mg/dL (maximum hypoglycemia risk); consequently, LBGI can theoretically assume values between 0 and 100 as well. Clinically relevant LBGI thresholds have been defined:
  1. LBGI <2.5: low hypoglycemia risk
  2. LBGI in 2.5-5: moderate hypoglycemia risk
  3. LBGI >5: high hypoglycemia risk.
Time Frame: 4 hours (dinner postprandial period); the final metric for each intervention type is obtained as the average over two consecutive camp days (days 1-2 for the first intervention; days 3-4 for the second intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard HCL Control - HCL Control With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control
Number analyzed (Participants) | 12 | 11
score on a scale
  Camp days 1-2 | 2.87 (2.59) | 3.19 (1.73)
  Camp days 3-4 | 1.1 (0.78) | 1.70 (0.79)
Statistical Analysis 1: Comparison: Standard HCL Control - HCL Control With Smart Bolus Calculator vs HCL Control With Smart Bolus Calculator - Standard HCL Control; The study followed a randomized crossover design, with two study groups and two intervention types; the two groups differed in the order they received the two intervention types. To test the hypothesis that "HCL Control with Smart Bolus Calculator" reduces exposure to hypoglycemia with respect to "Standard HCL Control", a mixed ANOVA was performed with LBGI as outcome measure, study group as between-subject factor, and intervention type as within-subject factor; Test type: Superiority; p = 0.733, ANOVA — For interaction between study group and intervention

2. Secondary Outcome: Percentage of Time Spent Below 70 mg/dL
Description: Percentage of CGM readings in hypoglycemia below 70 mg/dL
Time Frame: 4 hour (dinner postprandial period); average over two consecutive days for each intervention type, as described for primary outcome
Measure: Mean (Standard Deviation); unit: percentage of time spent below 70 mg/dL
Arm/Group | Standard HCL Control - HCL Control With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control
Number analyzed (Participants) | 12 | 11
percentage of time spent below 70 mg/dL
  Camp days 1-2 | 10.33 (14.55) | 12.08 (7.88)
  Camp days 3-4 | 2.31 (3.16) | 5.00 (3.61)
Statistical Analysis 1: Comparison: Standard HCL Control - HCL Control With Smart Bolus Calculator vs HCL Control With Smart Bolus Calculator - Standard HCL Control; The study followed a randomized crossover design, with two study groups and two intervention types; the two groups differed in the order they received the two intervention types. A mixed ANOVA was performed with percentage of time spent below 70 mg/dL as outcome measure, study group as between-subject factor, and intervention type as within-subject factor; Test type: Superiority; p = 0.824, ANOVA — For interaction between study group and intervention

3. Secondary Outcome: Percentage of Time Spent in 70-180 mg/dL
Description: Percentage of CGM readings in normoglycemia between 70-180 mg/dL
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time spent in 70-180 mg/dL
Arm/Group | Standard HCL Control - HCL Control With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control
Number analyzed (Participants) | 12 | 11
percentage of time spent in 70-180 mg/dL
  Camp days 1-2 | 83.16 (14.40) | 78.16 (20.98)
  Camp days 3-4 | 81.47 (15.30) | 85.44 (17.73)
Statistical Analysis 1: Comparison: Standard HCL Control - HCL Control With Smart Bolus Calculator; The study followed a randomized crossover design, with two study groups and two intervention types; the two groups differed in the order they received the two intervention types. A mixed ANOVA was performed with percentage of time spent in 70-180 mg/dL as outcome measure, study group as between-subject factor, and intervention type as within-subject factor; Test type: Superiority; p = 0.402, ANOVA — For interaction between study group and intervention

4. Secondary Outcome: Percentage of Time Spent Above 180 mg/dL
Description: Percentage of CGM readings in hyperglycemia above 180 mg/dL
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time spent above 180 mg/dL
Arm/Group | Standard HCL Control - HCL Control With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control
Number analyzed (Participants) | 12 | 11
percentage of time spent above 180 mg/dL
  Camp days 1-2 | 6.51 (9.69) | 9.76 (21.25)
  Camp days 3-4 | 16.22 (16.37) | 9.56 (17.63)
Statistical Analysis 1: Comparison: Standard HCL Control - HCL Control With Smart Bolus Calculator; The study followed a randomized crossover design, with two study groups and two intervention types; the two groups differed in the order they received the two intervention types. A mixed ANOVA was performed with percentage of time spent above 180 mg/dL as outcome measure, study group as between-subject factor, and intervention type as within-subject factor; Test type: Superiority; p = 0.300, ANOVA — For interaction between study group and intervention

5. Secondary Outcome: High Blood Glucose Index (HBGI)
Description: HBGI computed from CGM collected in the four hours following the dinner meal.
  HBGI is a metric quantifying the risk for hyperglycemia (the higher the HBGI, the higher the exposure to/risk of hyperglycemia), calculated based on the following two steps:
  1. Transforming each CGM reading in the time-series of length N into a hyperglycemia risk score (rH(i), i=1,...,N) by applying the following transformation:
     rH(i) = 10 x (1.509 x (log(CGM(i))^1.084 - 5.381))^2, if CGM(i) >112.5 mg/dL; rH(i) = 0, if CGM(i) <=112.5 mg/dL
  2. Averaging the risk scores rH(i), i=1,...,N.
  The hyperglycemia risk score ranges from 0 for CGM readings <=112.5 mg/dL (no hyperglycemia risk) to 100 for CGM readings =600 mg/dL (maximum hyperglycemia risk); consequently, HBGI can theoretically assume values between 0 and 100 as well. Clinically relevant HBGI thresholds have been defined:
  1. HBGI <4.5: low hyperglycemia risk
  2. HBGI in 4.5-9: moderate hyperglycemia risk
  3. HBGI >9: high hyperglycemia risk.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard HCL Control - HCL Control With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control
Number analyzed (Participants) | 12 | 11
score on a scale
  Camp days 1-2 | 1.64 (1.73) | 3.51 (8.45)
  Camp days 3-4 | 4.10 (4.74) | 1.85 (2.60)
Statistical Analysis 1: Comparison: Standard HCL Control - HCL Control With Smart Bolus Calculator vs HCL Control With Smart Bolus Calculator - Standard HCL Control; The study followed a randomized crossover design, with two study groups and two intervention types; the two groups differed in the order they received the two intervention types. A mixed ANOVA was performed with HBGI as outcome measure, study group as between-subject factor, and intervention type as within-subject factor; Test type: Superiority; p = 0.168, ANOVA — For interaction between study arm and intervention

6. Secondary Outcome: CGM Coefficient of Variation
Description: CGM coefficient of variation as a measure of glucose variability
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Standard HCL Control - HCL Control With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control
Number analyzed (Participants) | 12 | 11
percent
  Camp days 1-2 | 25.36 (5.81) | 25.74 (8.69)
  Camp days 3-4 | 24.01 (5.14) | 21.74 (5.81)
Statistical Analysis 1: Comparison: Standard HCL Control - HCL Control With Smart Bolus Calculator vs HCL Control With Smart Bolus Calculator - Standard HCL Control; The study followed a randomized crossover design, with two study groups and two intervention types; the two groups differed in the order they received the two intervention types. A mixed ANOVA was performed with CGM coefficient of variation as outcome measure, study group as between-subject factor, and intervention type as within-subject factor; Test type: Superiority; p = 0.476, ANOVA — For interaction between study group and intervention

7. Secondary Outcome: Total Amount of Carbohydrate Administered as Rescue Treatments
Description: Total amount of carbohydrate administered as rescue treatments per study protocol
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Standard HCL Control - HCL Control With Smart Bolus Calculator | HCL Control With Smart Bolus Calculator - Standard HCL Control
Number analyzed (Participants) | 12 | 11
grams
  Camp days 1-2 | 29.75 (25.11) | 37.45 (23.51)
  Camp days 3-4 | 11.54 (10.69) | 20.41 (14.56)
Statistical Analysis 1: Comparison: Standard HCL Control - HCL Control With Smart Bolus Calculator vs HCL Control With Smart Bolus Calculator - Standard HCL Control; The study followed a randomized crossover design, with two study groups and two intervention types; the two groups differed in the order they received the two intervention types. A mixed ANOVA was performed with total amount of carbohydrate administered as rescue treatments as outcome measure, study group as between-subject factor, and intervention type as within-subject factor; Test type: Superiority; p = 0.914, ANOVA — For interaction between study group and intervention

ADVERSE EVENTS:
Time Frame: About six months
Groups:
- Standard HCL Control: Use of standard HCL system
- HCL Control With Smart Bolus Calculator: Use of HCL system with smart bolus calculator informed by insulin sensitivity
Arm/Group | Standard HCL Control | HCL Control With Smart Bolus Calculator
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard HCL Control (N=25) | HCL Control With Smart Bolus Calculator (N=25)
Vomiting (General disorders) | 0 | 1
Sore Throat (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was a 4-day randomized crossover camp, with participants crossing from 1st to 2nd intervention at the end of day 2. Protocol imposed meals in days 1-2 to be repeated in days 3-4. However, meal carbohydrate content used for insulin dosing was reduced in days 3-4 because of suspicion of inaccurate carb estimate from the kitchen and to limit hypoglycemia. This led to significant hypoglycemia reduction in days 3-4, independently of the intervention phase, which complicates data interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04878120/Prot_SAP_000.pdf
  • Informed Consent Form: Minor Assent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04878120/ICF_001.pdf
  • Informed Consent Form: Minor Assent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04878120/ICF_002.pdf